CLINICAL TRIAL: NCT01596998
Title: Comparison of Plasma Concentrations of Levobupivacaine With and Without Epinephrine for Transversus Abdominis Plane Block Under Ultrasound.
Brief Title: Plasma Concentrations of Levobupivacaine With and Without Epinephrine in Transversus Abdominis Plane Blocks
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, Fernando Altermatt, Profesor Asistente, Departamento de Anestesiología, Pontificia Universidad Catolica de Chile
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 11-026
Record Dates: First submitted 2012-05-09; First posted 2012-05-11 (Estimated); Last update posted 2012-05-11 (Estimated); Status verified 2012-05

CONDITIONS: Transversus Abdominis Plane Block
Keywords: anesthesia, conduction; transversus abdominis plane block; Vasoconstrictor Agents; Ultrasonography
MeSH Terms: interventions — Levobupivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levobupivacaine without epinephrine (Active Comparator)
  Interventions: Drug: Levobupivacaine without epinephrine; Other: Monitoring; Other: Determining the extent of the block
- Levobupivacaine with epinephrine (Experimental)
  Interventions: Drug: Levobupivacaine with epinephrine; Other: Monitoring

INTERVENTIONS:
Drug: Levobupivacaine with epinephrine — The subjects were randomized to receive a unilateral TAP block. This was realized using a sterile technique, guided by ultrasound. Two operators with experience in ultrasound-guided regional blocks performed all procedures. A high-resolution linear U.S. transducer (L38x/10-5 MHz Sonosite M-Turbo®, Bothell, WA) and a Stimuplex 100 mm needle, 20 gauge (B. Braun Stimuplex, Melgusen, Germany) were used. After obtaining a clear view of the blocking plane, between internal oblique and transverse muscles, 20 ml of levobupivacaine 0.25% with 5 µg/mL epinephrine were injected.
  Arms: Levobupivacaine with epinephrine
Drug: Levobupivacaine without epinephrine — The subjects were randomized to receive a unilateral TAP block. This was realized using a sterile technique, guided by ultrasound. Two operators with experience in ultrasound-guided regional blocks performed all procedures. A high-resolution linear U.S. transducer (L38x/10-5 MHz, Sonosite M-Turbo ®, Bothell, WA) and a Stimuplex 100 mm needle, 20 gauge (B. Braun Stimuplex, Melgusen, Germany) were used. After obtaining a clear view of the blocking plane, between internal oblique and transverse muscles, 20 ml of levobupivacaine 0.25% were injected.
  Arms: Levobupivacaine without epinephrine
Other: Monitoring — Standard anesthetic monitoring was used, including continuous electrocardiogram, non invasive blood pressure and peripheral oxygen saturation. Later, under local anesthesia a permeable venous line and an arterial line were installed for blood sampling measures to determine local anesthetic plasma levels.
Other: Determining the extent of the block — The extent of sensory block was measured by assessment of temperature, soft and hard touch using alcohol, cotton and pin prick respectively. These measurements were made every 10 minutes during the first hour and every 30 minutes to complete 4 hours.
  Arms: Levobupivacaine without epinephrine

SUMMARY:
The aim of this study is to determine the effect of the addition of vasoconstrictor in the plasma concentrations achieved and the extent of the transversus abdominis plane block in healthy male volunteers.

DETAILED DESCRIPTION:
Use of TAP blocks, decreases use of opioids and reduces pain scores during the postoperative period after surgeries involving the anterior abdominal wall. However, the information regarding the sensitive range of the blockade and its duration is still limited. Since that the area of administration is an intermuscular plane, it is possible to infer a large area of absorption. Knowing plasma concentrations is essential to balance the usefulness of this technique with potential systemic toxicity associated with its use.

As an additional effect, clinically, the use of vasoconstrictors may prolong the duration of the blockade significantly, depending on the drug used and site of administration. To date, no studies evaluating the effect of the addition of vasoconstrictor both in the plasma concentrations achieved, and the quality, extent and duration of the TAP block.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers
* ASA I-II

Exclusion Criteria:

* BMI > 30kg m-2
* Patients with allergy to study drugs

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Effect of the addition of vasoconstrictor in the plasma concentrations achieved | Since the beginning of the block up to 90 minutes after

SECONDARY OUTCOMES:
Determine the mapping of sensory block in the abdominal wall after the completion of a U.S. guided TAP Block in healthy volunteers. | Since the beginning of the block up to 4 hours after

CONTACTS AND LOCATIONS:
Overall Officials: Fernando R Altermatt, MD, Principal Investigator — Departamento de Anestesiología, Hospital Clínico Pontificia Universidad Católica de Chile
Locations (1):
- Hospital Clinico Universidad Catolica, Santiago, Santiago Metropolitan, Chile